CLINICAL TRIAL: NCT00057993
Title: Phase II Study Of Herceptin And Exemestane For Treatment Of Postmenopausal Women With Metastatic Hormone-Responsive, HER2/NEU Positive Breast Cancer
Brief Title: Trastuzumab and Exemestane in Treating Postmenopausal Women With Metastatic or Locally Advanced Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to accrue subjects to the study after 2 years - closed per request by Data Monitoring Committee.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: NU 01B4; NU-01B4; PHARMACIA-NU-01B4
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: trastuzumab
Drug: exemestane

SUMMARY:
RATIONALE: The monoclonal antibody trastuzumab can locate breast cancer cells that have HER2 on their surface and either kill them or deliver tumor-killing substances to them without harming normal cells. Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using exemestane may fight breast cancer by reducing the production of estrogen. Combining trastuzumab with exemestane may be an effective treatment for breast cancer with high amounts of HER2.

PURPOSE: Phase II trial to study the effectiveness of combining trastuzumab with exemestane in treating postmenopausal women who have metastatic or locally advanced HER2-positive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of exemestane and trastuzumab (Herceptin), in terms of response rate and time to progression, in postmenopausal women with metastatic or locally advanced hormone-responsive, HER2/neu positive breast cancer.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive trastuzumab (Herceptin) IV over 30-90 minutes on day 1 and oral exemestane once daily. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 18-60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Stage IV or locally advanced disease

    * Staged by bone scan or CT scan of chest and/or abdomen within the past 6 weeks
* HER2/neu positive by fluorescent in situ hybridization (if 2+ by immunohistochemistry) or 3+ by immunohistochemistry
* Measurable disease defined by 1 of the following criteria:

  * At least 1 dimension at least 1 cm by CT scan or other imaging scan
  * At least 1 diameter at least 1 cm by plain x-ray (excluding bone lesions)
  * Palpable lesion with both diameters at least 1 cm with caliper OR
* Evaluable disease defined by 1 of the following criteria:

  * Positive bone scan
  * Palpable masses with diameter less than 1 cm, masses with margins not clearly defined on CT scan or x-ray, or with both diameters less than 1 cm
  * Bone scan and CA 27.29 if bone scan only evaluable disease
* Hormone receptor status:

  * Estrogen receptor and/or progesterone receptor positive

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Postmenopausal by 1 of the following criteria:

  * 60 years of age and over
  * 45 years of age and over with amenorrhea more than 12 months and an intact uterus
  * Follicle-stimulating hormone levels within postmenopausal range
  * Undergone bilateral oophorectomy

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin less than 1.5 times upper limit of normal

Renal

* Creatinine less than 2 mg/dL

Cardiovascular

* Ejection fraction greater than 50%

Other

* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior trastuzumab (Herceptin)

Chemotherapy

* Prior chemotherapy allowed

Endocrine therapy

* No prior exemestane
* No other prior hormonal agent (except tamoxifen)

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-07; Primary Completion 2004-08; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Virginia G. Kaklamani, MD, Principal Investigator — Robert H. Lurie Cancer Center